CLINICAL TRIAL: NCT00197925
Title: Vaccination With Autologous Dendritic Cells Pulsed With Onco-Peptides for Treatment of Patients With Metastatic Breast Cancer.A Phase I/II Study
Brief Title: Dendritic Cell Based Therapy of Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: all patients recruited
Sponsor: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA0415
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2008-01

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; dendritic cells; vaccine
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Biological: Onco-peptide loaded autologous dendritic cells

SUMMARY:
The study aim to show if vaccination with autologous dendritic cells pulsed with onco-peptides in combination with adjuvant cytokine can induce a measurable immune response in patients with metastatic breast cancer, and to evaluate the clinical effect (objective response rate) of the vaccination regime.

DETAILED DESCRIPTION:
HLA A2 positive patients are treated with PADRE and oncopeptide pulsed DC; p53, survivin and telomerase peptides. Each patient is given 6 immunizations with at least 5x106 peptide/lysate pulsed autologous DC. Vaccination 1-4 is given weekly and 4-6 at 2-week intervals. Those patients who exhibit stable disease, partial response or complete response after 6 injections will be given 4 more vaccinations at 2-week interval. The vaccine is applied by either intranodal or intradermal injection near the inguinal region. For adjuvant used IL-2 2 MIU sc. day 2-6. Scans and re-staging tests are performed at scheduled intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven progressive metastatic or locally advanced breast cancer
* No standard treatment indicated
* Age: > 18
* WHO-Performance Status 0-1
* At least tone measurable tumor lesions according to the RECIST criteria.
* Expression of the HLA-A2 tissue type
* Life expectancy more than 3 months
* Acceptable CBC and blood chemistry results
* Written informed consent

Exclusion Criteria:

* Patients with a history of any other neoplastic disease less than 5 years ago (excepting treated carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin).
* Patients with metastatic disease in the central nervous system (CNS).
* Patients with other significant illness including severe allergy, asthma, angina pectoris or congestive heart failure.
* Patients with acute or chronic infection including HIV, hepatitis and tuberculosis.
* Patients who are pregnant.
* Patients who have received antineoplastic therapy including chemotherapy or immunotherapy less than 4 weeks before beginning the trial.
* Patients who receive corticosteroids or other immunosuppressive agents.
* Patients with active autoimmune diseases such as lupus erythematosus, rheumatoid arthritis or thyroiditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-09

PRIMARY OUTCOMES:
Primary aim of the study is to evaluate tolerability and safety of the treatment.

SECONDARY OUTCOMES:
Secondary aims: evaluation of treatment induced immune response and clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, MD, PHD, Principal Investigator — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark
Locations (1):
- Department of Oncology, Herlev, Denmark

REFERENCES:
- [Background] Svane IM, Pedersen AE, Johnsen HE, Nielsen D, Kamby C, Gaarsdal E, Nikolajsen K, Buus S, Claesson MH. Vaccination with p53-peptide-pulsed dendritic cells, of patients with advanced breast cancer: report from a phase I study. Cancer Immunol Immunother. 2004 Jul;53(7):633-41. doi: 10.1007/s00262-003-0493-5. Epub 2004 Feb 25. PMID 14985857